CLINICAL TRIAL: NCT04718376
Title: A Multicenter, Open-label, Single-arm, Phase Ib Study to Evaluate the Safety and Efficacy of Mitoxantrone Hydrochloride Liposome Injection in Subjects With Platinum-Resistant or Platinum-Refractory Relapsed Ovarian Cancer
Brief Title: A Study of Mitoxantrone Hydrochloride Liposome Injection in the Treatment of Relapsed Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor has adjusted its R&D strategy.
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE071-CSP-015
Record Dates: First submitted 2020-12-14; First posted 2021-01-22 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2021-05

CONDITIONS: Platinum-resistant Ovarian Cancer
Keywords: platinum-refractory, platinum-resistant, ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Injections, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitoxantrone Hydrochloride Liposome Injection (Experimental): Subjects with Platinum-Resistant or Platinum-Refractory Relapsed Ovarian Cancer will receive 20 mg/m2 Mitoxantrone Hydrochloride Liposome every 21 days (a cycle) for a maximum of 8 cycles.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome, intravenous injection (IV)

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome, intravenous injection (IV) — All subjects will receive Mitoxantrone Hydrochloride Liposome 20 mg/m2, IV, on day 1 of each 21-day cycle (q3w).

SUMMARY:
This is a multicenter, open-label, single-arm, phase Ib study to evaluate the safety and efficacy of Mitoxantrone Hydrochloride Liposome in subjects with Platinum-Resistant or Platinum-Refractory Relapsed Ovarian Cancer.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm, phase Ib study to evaluate the safety and efficacy of Mitoxantrone Hydrochloride Liposome in subjects with Platinum-Resistant or Platinum-Refractory Relapsed Ovarian Cancer. At least 30 subjects will be recruited in this study. The subjects will receive Mitoxantrone Hydrochloride Liposome 20 mg/m2 by an intravenous infusion (IV), every 21 days (q3w, 1 cycle). All patients will receive the treatment until disease progression, intolerable toxic reaction, death, or withdrawal by investigator or patient decision (a maximum of 8 cycles). Delays in drug administration is allowed from the cycle 2, however, the delays should be no more than 3 weeks. Dose adjustments after the cycle 2 is permitted, and the minimum dose is 12mg/m2.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign informed consent;
2. Age ≥18, female;
3. Histologically confirmed diagnosis of epithelial ovarian cancer, fallopian tube carcinoma or primary peritoneal carcinoma (excluding low grade serous carcinoma and mucous carcinoma);
4. Fail to respond to or progressed on the standard platinum-based therapy ;
5. At least one measurable lesion according to RECIST v1.1;
6. ECOG performance status of 0 to 2;
7. Life expectancy ≥ 12 weeks;
8. AEs from the previous treatment have resolved to ≤ Grade 1 based on CTCAE (except for the toxicity without safety risk judged by the investigator, such as hair loss, hyperpigmentation);
9. Adequate organ function;
10. Subjects of childbearing potential must agree to use effective contraceptive measures. Female subjects must have a negative pregnancy test before enrolment;
11. Fully comply with the protocol.

Exclusion Criteria:

1. History of allergy to mitoxantrone hydrochloride or any excipients of the study drug;
2. Untreated or symptomatic central nervous system (CNS) metastases;
3. Pericardial effusion with clinical symptoms
4. History of allotransplantation;
5. Known hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) or other active viral infection;
6. Serious infection or interstitial pneumonia within 1 week prior to the first dose administration;
7. Use of other anticancer treatment within 4 weeks prior to the first dose administration;
8. Enrolled in any other clinical trials within 4 weeks prior to the first dose administration;
9. Major surgery within 3 months prior to the first dose administration, or have a surgical schedule during the study period;
10. Thrombosis or thromboembolism within 6 months prior to screening;
11. History of, or known additional malignant tumor within 3 years, except for tumors have been cured and have not recurred, and carcinoma in situ;
12. Impaired cardiac function or serious cardiac disease;
13. Previous treatment with adriamycin or other anthracyclines, and the total cumulative dose of prior adriamycin or equivalent is >350 mg/m2.
14. Pregnant or lactating female;
15. Serious and/or uncontrolled systemic diseases;
16. Not suitable for this study as decided by the investigator due to other reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
adverse events (AEs) | from the initiation of the first dose to 28 days after the last dose，assessed up to 36 months
  The incidence and severity of AEs, abnormalities in physical exams, vital sign assessments, clinical laboratory assessments, ultrasonic cardiograms (UCGs) and electrocardiographs (ECGs).

SECONDARY OUTCOMES:
overall response rate (ORR) | From the enrollment to the final documentation of response of the last subject (assessed up to 36 months)
  To investigate the preliminary antitumor efficacy
duration of response (DoR) | From the enrollment to death, lost to follow-up, withdrawal, or study end, whichever occurred first, assessed up to 36 months
  To investigate the preliminary antitumor efficacy
duration of complete response (DCR) | From the enrollment to death, lost to follow-up, withdrawal, or study end, whichever occurred first, assessed up to 36 months
  To investigate the preliminary antitumor efficacy
progression-free survival (PFS) | From the enrollment to death, lost to follow-up, withdrawal, or study end, whichever occurred first, assessed up to 36 months
  To investigate the preliminary antitumor efficacy
overall survival (OS) | From the enrollment to the death of last subject or the end of the clinical trial (assessed up to 36 months)
  To investigate the preliminary antitumor efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Qi Zhou, Master, Principal Investigator — Chongqing University Cancer Hospital
Locations (7):
- China (7):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Guizhou Cancer Hospital, Guiyang, Guizhou
  - Harbin Medical University Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No